CLINICAL TRIAL: NCT05745688
Title: Epidemiological Study on Gender Bias and Overtreatment in Primary Care Setting
Brief Title: Gender Bias and Overtreatment in Primary Care
Status: Completed | Type: Observational
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, José Joaquín Mira, Professor, Universidad Miguel Hernandez de Elche
Other Study IDs: OVERGEND Data
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Any Condition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to analyze if there are differences between men and women in the frequency of ignoring "Do not do" recommendations in primary care setting.

DETAILED DESCRIPTION:
First, using the Delphi technique, a consensus will be reached on those "Do Not Do" recommendations that should be included in the retrospective analysis study. The selection criteria for these recommendations will be if they are about pharmacological treatments, considered to persist in clinical practice in primary care, their relationship with factors associated with sex and gender, and if ignoring the "Do not do" recommendation could cause a serious adverse event.

Second, a retrospective cohort study will be carried out including patients who attended primary care consultation in Alicante from 1st January 2022 to 31st December 2022. Data source will be the electronic record management system of the autonomous community of Valencia (named ABUCASIS), and they will be provided by the Ambulatory Assistance Information System (SIA-GAIA). Investigators will analyze the frequency of ignoring the "Do not do" recommendations previously selected by consensus by sex and age range.

ELIGIBILITY:
Inclusion Criteria:

* Attending primary care consultation from 1 January 2022 to 31 December 2022.
* Adults

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults attending primary care consultation from 1 January 2022 to 31 December 2022
Sampling Method: Non-Probability Sample
Enrollment: 1048000 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Number of female patients who were recommended "do not do" | From 1st January 2022 to 31 December 2022
  Number of female patients who were recommended "do not do"
Number of male patients who were recommended "do not do" | From 1st January 2022 to 31 December 2022
  Number of male patients who were recommended "do not do"

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Juan de Alicante, Sant Joan d'Alacant, Alicante, Spain